CLINICAL TRIAL: NCT05275413
Title: Engaging the Whole Family to Support Expectant Mothers: A Family-based mHealth Intervention to Reduce Maternal Postnatal Depression and Promote Family Health
Brief Title: mHealth Intervention to Reduce Maternal Postnatal Depression and Promote Family Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Kwong Wah Hospital (Other); The University of Hong Kong (Other); University of Glasgow (Other); Tsan Yuk Hospital, Hong Kong (Unknown)
Responsible Party: Principal Investigator, Dr Camilla Lo, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KC/KE-20-0119/ER-2
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Postnatal Depression; Quality of Life; Family Relations
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- family-based mHealth intervention (Experimental): The expectant mothers and their family members (fathers and grandparents) in this group will receive health education and support and family support via a smartphone app.
  Interventions: Behavioral: family-based mHealth Intervention
- mother-only mHealth intervention (Experimental): The expectant mothers in this group will receive health education and support via a smartphone app.
  Interventions: Behavioral: mother-only mHealth Intervention
- Health education (Active Comparator): The expectant mothers in the control group will receive health education via a smartphone app.
  Interventions: Other: Health education

INTERVENTIONS:
Behavioral: family-based mHealth Intervention — The intervention consists of three versions: mother, father, and grandparent. The app consists of health information about pregnancy, postnatal care, and infant care in the form of brief texts and short videos. Each versions have their unique features, such as a platform to ask questions in mother version, a quiz game to promote fathers' knowledge related to father's involvement, educational materials tailored for grandparents. An obstetrician and a social worker will respond to the questions. Details please refer to the proposal.
  Arms: family-based mHealth intervention
Behavioral: mother-only mHealth Intervention — The expectant mothers in this group will receive information about pregnancy, postnatal care, and infant care in the form of brief texts and short videos via a smartphone app. The expectant mothers will also have access to a platform in the smartphone app to ask questions about their pregnancy. An obstetrician will respond to the questions.
  Arms: mother-only mHealth intervention
Other: Health education — The expectant mothers in the control group will receive information about pregnancy, postnatal care, and infant care in the form of brief texts and short videos via a smartphone app.
  Arms: Health education

SUMMARY:
The proposed study is to test the effectiveness of a culturally-attuned, family-based mobile health (mHealth) intervention in reducing symptoms of postnatal depression and promoting health among expectant mothers in Hong Kong. Using a family perspective, the proposed mHealth intervention will engage family members, including expectant fathers and grandparents, in providing support to expectant mothers. Expectant mothers and their family members will be recruited at antenatal clinics at two public hospitals in Hong Kong and randomized to receive the family-based mHealth intervention (experimental), the mother-only mHealth intervention (experimental), or the health education (control). Maternal depression, anxiety and stress, perceived social support, health-related quality of life, and perceived family cohesion will be assessed at recruitment and four weeks after childbirth. For family members, symptoms of anxiety and stress, health-related quality of life, and perceived family cohesion will be measured.

DETAILED DESCRIPTION:
Postnatal depression is a prevalent health issue affecting women. Although empirical evidence has proven the effectiveness of face-to-face antenatal classes in reducing perinatal distress, the availability of such support is often limited and is insufficient to benefit all parents who need it. Another challenge in pregnancy support is the difficulty to engage family members in providing support to expectant mothers. To address these limitations, the proposed project aims to develop and test the effectiveness of a family-based mobile health (mHealth) intervention, which will engage family members, including expectant fathers and grandparents to provide support to expectant mothers.

Specifically, the family-based mHealth intervention consists of a smartphone app with different versions designed for expectant mothers, fathers, and grandparents. The smartphone app will provide a user-friendly platform for users to receive psychoeducation materials related to pregnancy (e.g. antenatal care, postnatal care, and infant care) and an interactive forum for all users to ask questions related to pregnancy and family communication, which will be answered by health and social care professionals. To enhance family's engagement, we will also include other functions in the app to encourage communications among family members and enhance family cohesion. These functions include a platform for family members to send texts and share photos, and a shared schedule with alerts for dates related to pregnancy (e.g. appointments for antenatal check-ups and expected delivery date).

Using a randomized controlled design, the proposed study will evaluate the effectiveness of the family-based mHealth intervention in reducing maternal postnatal depression and promoting health in expectant mothers and their family members (expectant fathers and grandparents). The study will recruit 1,578 expectant mothers and their family members at the antenatal clinics at two selected public hospitals in Hong Kong. The participants will be randomized into three groups (i) family-based mHealth intervention; (ii) mother-only mHealth intervention; and (iii) health information control. Participants will be asked to complete a survey with question items related to their physical and mental health, perceived social support and family cohesion, at recruitment and four weeks after childbirth.

It is hypothesized that the family-based mHealth intervention is more effective in reducing symptoms of postnatal depression, promoting health of expectant mothers and their family members, and promoting family cohesion than the mother-only mHealth intervention and the control.

ELIGIBILITY:
Inclusion Criteria:

1. Expectant mothers (18 years old or above) attending the antenatal clinics at two public hospitals, Kwong Wah Hospital and Tsan Yuk Hospital in Hong Kong and their family members.
2. Possession of a smartphone and a personal email address for receiving and sending information relevant to the study.
3. Willing to accept the study arrangements.

Exclusion Criteria:

1. Not able to understand written or spoken Chinese.
2. Expectant mothers whose EPDS score is equal to or high than the cut-off score of 10.
3. Not willing or not able to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1578 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Postnatal depression symptoms | 24 weeks after start of intervention
  Symptoms of maternal depression at four weeks postpartum will be assessed with the validated Chinese version of the 10-item Edinburgh Postnatal Depression Scale (EPDS).

SECONDARY OUTCOMES:
Perceived social support levels of expectant mothers | 24 weeks after start of intervention
  Perceived social support levels of expectant mothers will be assessed with the Chinese version of the 12-item Multidimensional Scale of Perceived Social Support (MSPSS).
Anxiety and stress levels of all participants | 24 weeks after start of intervention
  Anxiety and stress levels of all participants (including the expectant mothers, fathers, and grandparents) will be assessed with the Anxiety and Stress subscales of the Chinese version of the Depression Anxiety Stress Scale (DASS21).
Health-related quality of life (QoL) of all participants | 24 weeks after start of intervention
  Health-related quality of life (QoL) of all participants will be measured with the validated Chinese version of the Short-form-12 Health survey (SF-12 v2), which consists of 12 items to be computed as two composite scores: physical component score and mental component score.
Perceived family cohesion levels of all participants | 24 weeks after start of intervention
  Perceived family cohesion levels of all participants will be assessed using the nine-item Family Cohesion subscale of the Chinese version of the Family Environment Scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Kwong Wah Hospital, Hong Kong
  - Tsan Yuk Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT05275413/Prot_SAP_000.pdf